CLINICAL TRIAL: NCT04339205
Title: Diffusion Imaging in Acute Auto-immune Encephalitis : a Cohort of 80 Patients
Brief Title: Diffusion Imaging in Acute Auto-immune Encephalitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Imaging study
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Auto-immune Encephalitis
Keywords: MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of every MRI at presentation of the symptoms and then over a period of 3 to 24 months if available. — The radiologist will analyze the MRI of patients with proved auto-immune encephalitis realized at presentation of the symptoms. If available, the following-up MRIs will also be analyzed.
  At each assessment, four MRI sequences will be studied : diffusion, T2-weighted, susceptibility sensitive sequences, and T1 weighted after contrast enhanced with gadolinium.
  The radiologist will analyse the signal abnormalities, their localisation and the trophicity of the brain.
  We will then correlate the following clinical data collected for patients : age, sex, clinical presentation, clinical evolution, and tumor associated or not.

SUMMARY:
The aim of this non randomised retrospective study is to investigate the imaging (MRI) of auto-immune encephalitis at presentation, especially in diffusion-weighted sequences.

Indeed, few series describe the MRI aspect of auto-immune at their beginning. Recognize early MRI abnormalities seen in auto-immune encephalitis could help reduce the time to positive diagnosis and improve the therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Auto-immune encephalitis proved by biological results (blood and/or CSF sample)

Exclusion Criteria:

* No MRI available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with auto-immune encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
MRI characterization, especially in Diffusion-weighted magnetic resonance imaging (DWI-MRI), of auto-immune encephalitis at presentation. | at following-up until 24 months
  The radiologist will analyze the MRI of patients with proved auto-immune encephalitis realized at presentation of the symptoms. If available, the following-up MRIs will also be analyzed.
  At each assessment, four MRI sequences will be studied : diffusion, T2-weighted, susceptibility sensitive sequences, and T1 weighted after contrast enhanced with gadolinium.
  The radiologist will analyse the signal abnormalities, their localisation and the trophicity of the brain.
  We will then correlate the following clinical data collected for patients : age, sex, clinical presentation, clinical evolution, and tumor associated or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No